CLINICAL TRIAL: NCT04995393
Title: Standardization of Infants Heel Warming Before Capillary Blood Sampling - a Randomized Controlled Study
Brief Title: Heel Warming Before Capillary Blood Sampling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kolding Sygehus (Other)
Collaborators: Region of Southern Denmark (Other); Development and Innovation Fund at Lillebaelt Hospital (Unknown); The Research Council for Sygehus Lillebælt (Unknown); Sygekassernes Helsefond (Other); The Biomedical Laboratory Scientist Education and Research Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: S-20200082
Record Dates: First submitted 2021-08-02; First posted 2021-08-09 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Blood Specimen Collection
Keywords: Blood Specimen Collection; Phlebotomy; Infant, Newborn; Heating; Heel; Pain
MeSH Terms: conditions — Pain | interventions — Heating

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Also masked: Biomedical Laboratory Scientist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glove (Active Comparator): A heated glove containing water.
  Interventions: Procedure: Heating with a disposable glove containing water
- Blanket (Active Comparator): A heated blanket.
  Interventions: Procedure: Heating with a blanket
- Gel pack (Active Comparator): A heated gel pack.
  Interventions: Procedure: Heating with a gel pack

INTERVENTIONS:
Procedure: Heating with a disposable glove containing water — Heating of the infants heel with a glove before blood sampling.
  Arms: Glove
Procedure: Heating with a blanket — Heating of the infants heel with a blanket before blood sampling.
  Arms: Blanket
Procedure: Heating with a gel pack — Heating of the infants heel with a gel pack before blood sampling.
  Arms: Gel pack

SUMMARY:
Capillary blood sampling from the heel is often used in the treatment of infants admitted to neonatal intensive care (NICU). In Danish NICUs a heated blanket, a heated gel pad or a disposable glove with warm water are the methods most often used.

The purpose of this randomized controlled study is to investigate which of the mentioned heating methods ensures the best quality of the blood sample and provides the most gentle blood sampling for the infant.

DETAILED DESCRIPTION:
Some infants experience a difficult and painful blood sampling which can lead to bruised or swollen heels and a blood sample of poor quality. To minimize the risk of that, the infant's heel is heated before the procedure as described in standard GP42-A6 from The Clinical and Laboratory Standards Institute. However, no consensus exists on which heating method to use. The aim of this study is to compare three different heating methods in terms of which method can help reduce pain experienced by infants as well as increase the quality of the blood samples.

Infants (postmenstrual age ≥ 28 + 0) admitted to the NICU, Kolding Hospital and having a blood sample taken by a Biomedical Laboratory Scientist are invited to participate. A parental informed concent must be signed by both parents before participation.

Infants are randomized to one of the three heating methods: glove, blanket or gel pad.

The following blood sampling procedure is closely monitored to register data corresponding to the five outcome measures.

Furthermore the infants personal data, location of the infant during the procedure, surface temperature of the heel before and after heating, volume of sampled blood, sign of bruises and swelling as well as hematocrit are registered.

Data registration, web-based block randomization, data storage and statistical analysis are supported by OPEN (Open Patient data Explorative Network, University of Southern Denmark).

The study is registered as public research at the Region of Southern Denmark (journal no. 20/1316) and is approved by The Regional Committees on Health Research Ethics for Southern Denmark (ID S-20200082).

ELIGIBILITY:
Inclusion Criteria:

* PMA (postmenstrual age) ≥ 28+0
* Blood sampling performed by a Biomedical Laboratory Scientist

Exclusion Criteria:

* GA (gestational age) ≥ 44+0
* Weight > 6000 g
* Coagulation related disorder
* Severe illness/disorder
* Heel is bruised or swollen
* Parents not understanding written Danish language

Ages: 2 Hours to 77 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 176 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

PRIMARY OUTCOMES:
Speed of blood sampling | 10 minutes
  µl blood/sec
Duration of blood sampling | 10 minutes
  Sec

SECONDARY OUTCOMES:
Hemolysis index for potassium of the blood sample | 2 hours
Degree of squeezing the infants foot during blood sampling | 1 minute
  Scale 1 to 5
Number of heel punctures required to obtain the blood sample | 10 minutes
  1, 2, 3 or 4
ComfortNeo score of the infant during the blood sampling | 20 minutes
  Pain assessment COMFORTneo score - range is 6 to 30.

CONTACTS AND LOCATIONS:
Overall Officials: Jonna Skov Madsen, Study Director — Clinical Biochemistry and Immunology, Lillebaelt Hospital, University Hospital of Southern Denmark; Patricia Diana Soerensen, Study Chair — Clinical Biochemistry and Immunology, Lillebaelt Hospital, University Hospital of Southern Denmark; Ulla List Toennesen, Principal Investigator — Clinical Biochemistry and Immunology, Lillebaelt Hospital, University Hospital of Southern Denmark
Locations (1):
- Neonatal intensive care (NICU), Lillebaelt Hospital, University Hospital of Southern Denmark, Kolding, Region Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valeri BO, Holsti L, Linhares MB. Neonatal pain and developmental outcomes in children born preterm: a systematic review. Clin J Pain. 2015 Apr;31(4):355-62. doi: 10.1097/AJP.0000000000000114. PMID 24866853
- [Background] Anand KJ; International Evidence-Based Group for Neonatal Pain. Consensus statement for the prevention and management of pain in the newborn. Arch Pediatr Adolesc Med. 2001 Feb;155(2):173-80. doi: 10.1001/archpedi.155.2.173. PMID 11177093
- [Background] Losacco V, Cuttini M, Greisen G, Haumont D, Pallas-Alonso CR, Pierrat V, Warren I, Smit BJ, Westrup B, Sizun J; ESF Network. Heel blood sampling in European neonatal intensive care units: compliance with pain management guidelines. Arch Dis Child Fetal Neonatal Ed. 2011 Jan;96(1):F65-8. doi: 10.1136/adc.2010.186429. PMID 21177753
- [Background] Janes M, Pinelli J, Landry S, Downey S, Paes B. Comparison of capillary blood sampling using an automated incision device with and without warming the heel. J Perinatol. 2002 Mar;22(2):154-8. doi: 10.1038/sj.jp.7210583. PMID 11896522
- [Background] Aydin D, Inal S. Effects of breastfeeding and heel warming on pain levels during heel stick in neonates. Int J Nurs Pract. 2019 Jun;25(3):e12734. doi: 10.1111/ijn.12734. Epub 2019 Apr 17. PMID 30993840
- [Background] WHO Guidelines on Drawing Blood: Best Practices in Phlebotomy. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK138650/ PMID 23741774
- [Background] Hassan Z, Shah M. Scald injury from the Guthrie test: should the heel be warmed? Arch Dis Child Fetal Neonatal Ed. 2005 Nov;90(6):F533-4. doi: 10.1136/adc.2005.072678. PMID 16244215
- [Background] Shu SH, Lee YL, Hayter M, Wang RH. Efficacy of swaddling and heel warming on pain response to heel stick in neonates: a randomised control trial. J Clin Nurs. 2014 Nov;23(21-22):3107-14. doi: 10.1111/jocn.12549. Epub 2014 Jan 30. PMID 24476226
- [Background] Folk LA. Guide to capillary heelstick blood sampling in infants. Adv Neonatal Care. 2007 Aug;7(4):171-8. doi: 10.1097/01.ANC.0000286333.67928.04. PMID 17700190
- [Background] Sorrentino G, Fumagalli M, Milani S, Cortinovis I, Zorz A, Cavallaro G, Mosca F, Plevani L. The impact of automatic devices for capillary blood collection on efficiency and pain response in newborns: A randomized controlled trial. Int J Nurs Stud. 2017 Jul;72:24-29. doi: 10.1016/j.ijnurstu.2017.04.001. Epub 2017 Apr 11. PMID 28431226